CLINICAL TRIAL: NCT02907879
Title: Contrast Enhanced Ultrasound Imaging for Cerebral Perfusion Measurement in Cerebral Vasospasm After Subarachnoid Hemorrhage
Brief Title: Contrast Enhanced Ultrasound Imaging for Cerebral Perfusion Measurement in Cerebral Vasospasm After SAH
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SONO SAB
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage; Ultrasound perfusion imaging; cerebral hypoperfusion; vasospasm; DIND; infarction
MeSH Terms: conditions — Subarachnoid Hemorrhage; Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound perfusion imaging: Measuring methods of UPI with phase inversion harmonic imaging

SUMMARY:
The objective of the study is to assess brain tissue perfusion by ultrasound perfusion imaging. Specifically

* to diagnose brain tissue hypoperfusion due to CVS with contrast enhanced UPI and to assess specificity and sensitivity, and predictive values for detection of brain tissue hypoperfusion leading to infarction
* to test whether treatment-effects by induced hypertension, balloon-dilatation, or intra-arterial nimodipine infusion can be detected and quantified by UPI

DETAILED DESCRIPTION:
The aim of the study is to assess brain tissue perfusion by ultrasound perfusion imaging (UPI).

The specific aim is to diagnose brain tissue hypoperfusion leading to infarction due to CVS with ultrasound perfusion imaging (UPI) and to correlate it with the gold standard of diagnosis of brain infarcts, i.e. with MRI and CT. According to contrast enhanced UPI brain tissue will be classified as (1) normal, i.e. not leading to tissue infarction, (2) as hypoperfused, i.e. functionally impaired and prone to DIND and to infarction, or (3) non-perfused. Thus, temporary hypoperfusion that may be resolved by therapy or spontaneously, not leading to tissue infarction shall be assessed. This strategy will lead to guiding therapy by UPI.

Questionnaire:

* to assess cerebral perfusion in patients with SAH by contrast enhanced UPI
* to assess specificity and sensitivity, as well as positive and negative predictive values of contrast enhanced UPI for detection of brain tissue misery perfusion leading to infarction
* to evaluate feasibility and practicability of repeated bed-side assessments of UPI
* to test whether treatment-effects like induced hypertension, balloon-dilation, or intra-arterial nimodipine infusion can be detected and quantified by contrast enhanced UPI
* to analyze whether TCD or contrast enhanced UPI is superior for screening of CVS and detection of cerebral infarcts (vessel vs. tissue assessment)
* to correlate contrast enhanced UPI with perfusion measurements by CT-perfusion imaging

Ultrasound perfusion imaging (UPI) is able to detect cerebral hypoperfusion that can result in cerebral infarction in a clinical setting. As reference the incidence of cerebral infarcts is assessed by CT- and MR-imaging and cerebral perfusion is analyzed by CT-perfusion (CTP) imaging.

The day of the ictus (SAH) is defined as day 0. The ultrasound examinations will be performed at

* Day 0-4: one baseline UPI study will be performed. This time period (0-4) is set as baseline, because this baseline investigation will be performed before vasospasm develops. The current policy of early aneurysm treatment results in clipping or coiling of patients within 24-48 hours. The relevant phase of CVS, however, starts on day 4 to 5 after the ictus. The already established routine protocol with early CT and CTP imaging after aneurysm treatment allows differentiation between infarcts due to the procedure of aneurysm clipping or coiling, bleeding, edema, or surgical contusions from cerebral infarcts due to CVS that develop later on. This early routine CT imaging includes a CT-perfusion study on post-op day 1, serving as reference for the ultrasound perfusion measurements.
* Day 5-14: during the term with the highest risk for CVS, a UPI study will be performed every second day.
* Several events trigger additional UPI studies:

  * angiography (scheduled or emergency)
  * endovascular intervention (angioplasty or intraarterial nimodipine infusion)
  * CT or MRI study with new infarcts
  * Development of DIND or reversal of DIND
  * in case of placement of an intracerebral microprobe (rCBF or ptiO2) an UPI study will be performed when significant changes (rCBF drop below 20ml/100g/min or below 60% of baseline, ptiO2 drop below 10mmHg or below 60% of baseline) occur.

Currently all patients are scanned by MRI and or CT several times in the course of the disease. Each imaging study serves as reference for UPI.

During day 5-14 high risk patients (Fisher grade 3, or TCD > 150 cm/sec, or new deficit) receive one CT-perfusion study between day 7 and 11 (period of highest risk).

During day 5-14 patients with proven CVS (angiography) will receive two CT-perfusion studies, one at day 7, and one at day 11, or at the time when new deficits or infarcts evolve. Additional about 20% of patients will get MRI including perfusion weighted imaging (PWI). In these patients misery perfusion as detected by PWI serves as reference for UPI.

The actual UPI measurement takes place at the bedside, is performed by the study physician, and takes about 15 -30 minutes.

The trial duration per patient is 14 days during the initial hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Proven SAH (CT or lumbar puncture)
* Proven aneurysm (digital subtraction angiography or CT-angiography)
* Age >18
* Informed consent of patient or relative

Exclusion Criteria:

* Pregnancy and breast feeding
* Acute coronary syndromes, severe ischemic heart disease (requiring revascularisation), severe aortic and mitral valve disease, severe congestive heart failure (NYHA >III/IV)
* Severe pulmonary or renal dysfunction
* Known allergy or adverse reaction to contrast material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with aneurysmal SAH admitted to the Departments of Neurosurgery, Neurology, or Intensive Care Medicine, will be screened for enrollment in the study
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Detection of cerebral hypoperfusion leading to either infarcts, neurological deficits, or initiation of rescue therapy | 14 days after ictus
  (1) normal, i.e. with a perfusion delay < 2 sec, (2) hypoperfusion, i.e. with a perfusion delay ≥ 2sec and < 6 sec, and (3) no perfusion, i.e. with a perfusion delay ≥ 6 sec as compared with the average of the 2 thalamic territories of the unaffected side

SECONDARY OUTCOMES:
Correlation between UPI parameters and cerebral perfusion as assessed by CT-perfusion | Within 14 days after ictus
Correlation between UPI parameters and cerebral perfusion as assessed by MRI-perfusion | Within 14 days after ictus
Correlation between UPI parameters and flow velocities in the middle cerebral artery as measured by TCD | Within 14 days after ictus
Correlation between UPI parameters with vessel diameters of the MCA as assessed by DSA | Within 14 days after ictus

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Beck, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of Neurosurgery, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Reitmeir R, Eyding J, Oertel MF, Wiest R, Gralla J, Fischer U, Giquel PY, Weber S, Raabe A, Mattle HP, Z'Graggen WJ, Beck J. Is ultrasound perfusion imaging capable of detecting mismatch? A proof-of-concept study in acute stroke patients. J Cereb Blood Flow Metab. 2017 Apr;37(4):1517-1526. doi: 10.1177/0271678X16657574. Epub 2016 Jan 1. PMID 27389180
- [Background] de Rooij NK, Linn FH, van der Plas JA, Algra A, Rinkel GJ. Incidence of subarachnoid haemorrhage: a systematic review with emphasis on region, age, gender and time trends. J Neurol Neurosurg Psychiatry. 2007 Dec;78(12):1365-72. doi: 10.1136/jnnp.2007.117655. Epub 2007 Apr 30. PMID 17470467
- [Background] Feigin VL, Lawes CM, Bennett DA, Barker-Collo SL, Parag V. Worldwide stroke incidence and early case fatality reported in 56 population-based studies: a systematic review. Lancet Neurol. 2009 Apr;8(4):355-69. doi: 10.1016/S1474-4422(09)70025-0. Epub 2009 Feb 21. PMID 19233729
- [Background] Johnston SC, Selvin S, Gress DR. The burden, trends, and demographics of mortality from subarachnoid hemorrhage. Neurology. 1998 May;50(5):1413-8. doi: 10.1212/wnl.50.5.1413. PMID 9595997
- [Background] Weidauer S, Lanfermann H, Raabe A, Zanella F, Seifert V, Beck J. Impairment of cerebral perfusion and infarct patterns attributable to vasospasm after aneurysmal subarachnoid hemorrhage: a prospective MRI and DSA study. Stroke. 2007 Jun;38(6):1831-6. doi: 10.1161/STROKEAHA.106.477976. Epub 2007 Apr 19. PMID 17446425
- [Background] Vergouwen MD, Vermeulen M, Roos YB. Effect of nimodipine on outcome in patients with traumatic subarachnoid haemorrhage: a systematic review. Lancet Neurol. 2006 Dec;5(12):1029-32. doi: 10.1016/S1474-4422(06)70582-8. PMID 17110283
- [Background] Raabe A, Beck J, Keller M, Vatter H, Zimmermann M, Seifert V. Relative importance of hypertension compared with hypervolemia for increasing cerebral oxygenation in patients with cerebral vasospasm after subarachnoid hemorrhage. J Neurosurg. 2005 Dec;103(6):974-81. doi: 10.3171/jns.2005.103.6.0974. PMID 16381183
- [Background] Aaslid R, Huber P, Nornes H. Evaluation of cerebrovascular spasm with transcranial Doppler ultrasound. J Neurosurg. 1984 Jan;60(1):37-41. doi: 10.3171/jns.1984.60.1.0037. PMID 6689726
- [Background] Beck J, Raabe A, Lanfermann H, Seifert V, Weidauer S. Tissue at risk concept for endovascular treatment of severe vasospasm after aneurysmal subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1779-81. doi: 10.1136/jnnp.2004.036921. PMID 15548506
- [Background] Beck J, Raabe A, Lanfermann H, Seifert V, Weidauer S. Perfusion-weighted magnetic resonance imaging in patients with vasospasm: a useful new tool in the management of patients with subarachnoid hemorrhage. Neurosurgery. 2006 Mar;58(3):E590; author reply E590. doi: 10.1227/01.NEU.0000207963.98939.7B. No abstract available. PMID 16528172
- [Background] Eyding J, Krogias C, Schollhammer M, Eyding D, Wilkening W, Meves S, Schroder A, Przuntek H, Postert T. Contrast-enhanced ultrasonic parametric perfusion imaging detects dysfunctional tissue at risk in acute MCA stroke. J Cereb Blood Flow Metab. 2006 Apr;26(4):576-82. doi: 10.1038/sj.jcbfm.9600216. PMID 16121127
- [Background] Seidel G, Meyer-Wiethe K, Berdien G, Hollstein D, Toth D, Aach T. Ultrasound perfusion imaging in acute middle cerebral artery infarction predicts outcome. Stroke. 2004 May;35(5):1107-11. doi: 10.1161/01.STR.0000124125.19773.40. Epub 2004 Mar 18. PMID 15031454
- [Derived] Chapman F, Morrissey R, McDermott S, Cahours X, Verron T, Taverner V, Stevenson M, Nahde T. Evaluation of high-nicotine oral products shows potential to reduce tobacco-related harm by offering satisfying alternatives. Sci Rep. 2025 Oct 3;15(1):34636. doi: 10.1038/s41598-025-21812-x. PMID 41044396
- [Derived] Fung C, Heiland DH, Reitmeir R, Niesen WD, Raabe A, Eyding J, Schnell O, Rolz R, Z Graggen WJ, Beck J. Ultrasound Perfusion Imaging for the Detection of Cerebral Hypoperfusion After Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2022 Aug;37(1):149-159. doi: 10.1007/s12028-022-01460-z. Epub 2022 Feb 24. PMID 35211837